CLINICAL TRIAL: NCT05575193
Title: The Effect of Acupressure on Uremic Pruritus and Sleep Quality Among Patients Receiving Hemodialysis
Brief Title: Acupressure on Uremic Pruritus and Sleep Quality Among Patients Receiving Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, RN, DNSc, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202102EM001
Record Dates: First submitted 2022-09-28; First posted 2022-10-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hemodialysis; Uremic Pruritus
Keywords: Hemodialysis; Acupressure; Uremic Pruritus; Sleep Quality; Effect
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The patients receiving the intervention of acupressure are in the experimental group, while those who do not receive it are in the control group. The experimental group will receive the acupressure at the hemodialysis center for a total of 12 weeks, three times a week. The patients will receive 4 acupuncture points, including Quchi acupoint, Xuehai acupoint, Sanyinjiao acupoint, and Zusanli acupoint. Each acupoint will be pressed for 3 minutes, and totally 4 acupuncture points are 12 minutes. The effectiveness will be evaluated at the fourth week, eighth week and twelfth week. The effectiveness assessment in the study will use the "Visual Analog Scale (VAS)", "5D Pruritus Scale", and "Pittsburgh Sleep Quality Scale".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Group (Experimental): The patients receiving the intervention of acupressure are in the experimental group.The experimental group will receive the acupressure at the hemodialysis center for a total of 12 weeks, three times a week. The patients will receive 4 acupuncture points, including Quchi acupoint, Xuehai acupoint, Sanyinjiao acupoint, and Zusanli acupoint. Each acupoint will be pressed for 3 minutes, and totally 4 acupuncture points are 12 minutes. The effectiveness will be evaluated at the fourth week, eighth week and twelfth week.
  Interventions: Other: Acupressure
- Non-Acupressure Group (No Intervention): Acupressure is not provided, only general routines are performed. Pre-test and 3 post-tests of "Visual Analog Scale (VAS)", "5D Tickling Scale", and "Pittsburgh Sleep Quality Scale" are also required (week 4, week 8 and week 12).

INTERVENTIONS:
Other: Acupressure — The patients will receive 4 acupuncture points, including Quchi acupoint, Xuehai acupoint, Sanyinjiao acupoint, and Zusanli acupoint. Each acupoint will be pressed for 3 minutes, and totally 4 acupuncture points are 12 minutes.
  Arms: Acupressure Group

SUMMARY:
The research is to explore the effect of acupressure on uremic pruritus and sleep quality among patients receiving hemodialysis. The research method adopts the experimental research method using randomization. The patients receiving the intervention of acupressure are in the experimental group, while those who do not receive it are in the control group.

DETAILED DESCRIPTION:
There are about 60-90% of hemodialysis patients complain of itchy skin, which can cause the sleep quality decline. The important issue of non-invasive acupressure methods to relieve skin itching symptoms and to improve sleep quality are worth explored. Therefore, the research is to explore the effect of acupressure on uremic pruritus and sleep quality among patients receiving hemodialysis. The research method adopts the experimental research method using randomization. The patients receiving the intervention of acupressure are in the experimental group, while those who do not receive it are in the control group. The experimental group will receive the acupressure at the hemodialysis center for a total of 12 weeks, three times a week. The patients will receive 4 acupuncture points, including Quchi acupoint, Xuehai acupoint, Sanyinjiao acupoint, and Zusanli acupoint. Each acupoint will be pressed for 3 minutes, and totally 4 acupuncture points are 12 minutes. The effectiveness will be evaluated at the fourth week, eighth week and twelfth week. The effectiveness assessment in the study will use the "Visual Analog Scale (VAS)", "5D Pruritus Scale", and "Pittsburgh Sleep Quality Scale". This study uses the pre-test before the implementation of acupuncture, and uses the post-test at week 4, 8, and 12 end of acupuncture. Hopefully, this study may develop a beneficial non-drug care measures to improve the itching symptoms and sleep quality of hemodialysis patients, and to improve their quality of life. If this research result proves that the application of acupressure can be effective, it can not only improve the symptoms of itchy skin and sleep problems in hemodialysis patients, but also hope that can be extended to patients with end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

1. At least 3 months hemodialysis
2. At least 1 month have itching
3. At least mild itching on the 5D tickling scale (9-11 points)
4. Can answer questions correctly

Exclusion Criteria:

1. Skin-related disease
2. Liver disease
3. Psychiatric disorder
4. Cancer undergoing chemotherapy or radiation therapy
5. Nerve or vascular or soft tissue diseases of the extremitie
6. Infections or surgeries on the extremitie

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Pre-test
  The scale contains seven indicators (subjective sleep quality, sleep lag period, total sleep hours, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction). Each indicator has its own special scoring method. Indicators are calculated on a scale of 0-3, with a total score ranging from 0-21. The total score of the seven indicators is more than 5 points, the quality of sleep is poor, and the score is less than 5 points, the quality of sleep is good, which means that the higher the score, the worse the quality of sleep.
Pittsburgh Sleep Quality Index | Post-test at week 4
  The scale contains seven indicators (subjective sleep quality, sleep lag period, total sleep hours, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction). Each indicator has its own special scoring method. Indicators are calculated on a scale of 0-3, with a total score ranging from 0-21. The total score of the seven indicators is more than 5 points, the quality of sleep is poor, and the score is less than 5 points, the quality of sleep is good, which means that the higher the score, the worse the quality of sleep.
Pittsburgh Sleep Quality Index | Post-test at week 8
  The scale contains seven indicators (subjective sleep quality, sleep lag period, total sleep hours, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction). Each indicator has its own special scoring method. Indicators are calculated on a scale of 0-3, with a total score ranging from 0-21. The total score of the seven indicators is more than 5 points, the quality of sleep is poor, and the score is less than 5 points, the quality of sleep is good, which means that the higher the score, the worse the quality of sleep.
Pittsburgh Sleep Quality Index | Post-test at week 12
  The scale contains seven indicators (subjective sleep quality, sleep lag period, total sleep hours, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction). Each indicator has its own special scoring method. Indicators are calculated on a scale of 0-3, with a total score ranging from 0-21. The total score of the seven indicators is more than 5 points, the quality of sleep is poor, and the score is less than 5 points, the quality of sleep is good, which means that the higher the score, the worse the quality of sleep.
Visual analogue scale | Pre-test
  Is a subjective feeling, no itching = 0, very intense itching = 10, mainly to assess the intensity of the itching
Visual analogue scale | Post-test at week 4
  Is a subjective feeling, no itching = 0, very intense itching = 10, mainly to assess the intensity of the itching
Visual analogue scale | Post-test at week 8
  Is a subjective feeling, no itching = 0, very intense itching = 10, mainly to assess the intensity of the itching
Visual analogue scale | Post-test at week 12
  Is a subjective feeling, no itching = 0, very intense itching = 10, mainly to assess the intensity of the itching
5D Pruritus Scale | Pre-test
  It includes five items to assess: duration of tickling, degree of tickling, changes in tickling, effects of tickling on daily life (sleep, rest/social activities, housework/going out, work/class), and distribution of tickling, and the five items add up to a 5D tickling scale score, with a minimum of 5 points and a maximum of 25 points. Graded degree of itching: no tickling (≤ 8), mild tickling (9-11), moderate tickling (12-17), severe tickling (18-21), very severe itching (≥22)
5D Pruritus Scale | Post-test at week 4
  It includes five items to assess: duration of tickling, degree of tickling, changes in tickling, effects of tickling on daily life (sleep, rest/social activities, housework/going out, work/class), and distribution of tickling, and the five items add up to a 5D tickling scale score, with a minimum of 5 points and a maximum of 25 points. Graded degree of itching: no tickling (≤ 8), mild tickling (9-11), moderate tickling (12-17), severe tickling (18-21), very severe itching (≥22)
5D Pruritus Scale | Post-test at week 8
  It includes five items to assess: duration of tickling, degree of tickling, changes in tickling, effects of tickling on daily life (sleep, rest/social activities, housework/going out, work/class), and distribution of tickling, and the five items add up to a 5D tickling scale score, with a minimum of 5 points and a maximum of 25 points. Graded degree of itching: no tickling (≤ 8), mild tickling (9-11), moderate tickling (12-17), severe tickling (18-21), very severe itching (≥22)
5D Pruritus Scale | Post-test at week 12
  It includes five items to assess: duration of tickling, degree of tickling, changes in tickling, effects of tickling on daily life (sleep, rest/social activities, housework/going out, work/class), and distribution of tickling, and the five items add up to a 5D tickling scale score, with a minimum of 5 points and a maximum of 25 points. Graded degree of itching: no tickling (≤ 8), mild tickling (9-11), moderate tickling (12-17), severe tickling (18-21), very severe itching (≥22)

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Xuan-Yi Huang, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Che-Yi C, Wen CY, Min-Tsung K, Chiu-Ching H. Acupuncture in haemodialysis patients at the Quchi (LI11) acupoint for refractory uraemic pruritus. Nephrol Dial Transplant. 2005 Sep;20(9):1912-5. doi: 10.1093/ndt/gfh955. Epub 2005 Jun 28. PMID 15985509
- [Background] Badiee Aval S, Ravanshad Y, Azarfar A, Mehrad-Majd H, Torabi S, Ravanshad S. A Systematic Review and Meta-analysis of Using Acupuncture and Acupressure for Uremic Pruritus. Iran J Kidney Dis. 2018 Mar;12(2):78-83. PMID 29507269
- [Background] Kilic Akca N, Tasci S, Karatas N. Effect of acupressure on patients in Turkey receiving hemodialysis treatment for uremic pruritus. Altern Ther Health Med. 2013 Sep-Oct;19(5):12-8. PMID 23981400
- [Background] Kilic Akca N, Tasci S. Acupressure and Transcutaneous Electrical Acupoint Stimulation for Improving Uremic Pruritus: A Randomized, Controlled Trial. Altern Ther Health Med. 2016 Mar;22(3):18-24. PMID 27228268
- [Background] Karjalian F, Momennasab M, Yoosefinejad AK, Jahromi SE. The Effect of Acupressure on the Severity of Pruritus and Laboratory Parameters in Patients Undergoing Hemodialysis: A Randomized Clinical Trial. J Acupunct Meridian Stud. 2020 Aug;13(4):117-123. doi: 10.1016/j.jams.2020.05.002. Epub 2020 Jun 1. PMID 32497714
- [Background] Yan CN, Yao WG, Bao YJ, Shi XJ, Yu H, Yin PH, Liu GZ. Effect of Auricular Acupressure on Uremic Pruritus in Patients Receiving Hemodialysis Treatment: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2015;2015:593196. doi: 10.1155/2015/593196. Epub 2015 Oct 1. PMID 26495017